CLINICAL TRIAL: NCT03983551
Title: Comparing the Effect of Dipeptidyl-peptidase 4 Inhibitors and Sulfonylureas on Urinary Albumin Excretion in People With Type 2 Diabetes Mellitus
Brief Title: Comparing the Renal Effect of Dipeptidyl-peptidase 4 Inhibitors and Sulfonylureas
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Changhua Christian Hospital (Other)
Responsible Party: Principal Investigator, Po-Chung Cheng, Principal Investigator, Changhua Christian Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 190512
Record Dates: First submitted 2019-06-11; First posted 2019-06-12 (Actual); Last update posted 2019-06-14 (Actual); Status verified 2019-06

CONDITIONS: Type 2 Diabetes Mellitus; Proteinuria
Keywords: Type 2 diabetes mellitus; dipeptidyl peptidase 4 inhibitors; sulfonylureas; proteinuria
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Proteinuria | interventions — Dipeptidyl-Peptidase IV Inhibitors; Sulfonylurea Compounds

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dipeptidyl peptidase 4 inhibitors (Experimental): Vildagliptin 50 milligrams twice daily in addition to metformin 1000 milligrams once daily
  Interventions: Drug: Dipeptidyl Peptidase 4 Inhibitor
- Sulfonylureas (Active Comparator): Glimepiride 2 milligrams twice daily in addition to metformin 1000 milligrams once daily
  Interventions: Drug: Sulfonylurea

INTERVENTIONS:
Drug: Dipeptidyl Peptidase 4 Inhibitor — Vildagliptin 50 milligrams twice daily in addition to metformin 1000 milligrams once daily
  Other Names: DPP-4 inhibitor
  Arms: Dipeptidyl peptidase 4 inhibitors
Drug: Sulfonylurea — Glimepiride 2 milligrams twice daily in addition to metformin 1000 milligrams once daily
  Other Names: SU
  Arms: Sulfonylureas

SUMMARY:
Dipeptidyl peptidase 4 (DPP-4) inhibitors and sulfonylureas have been extensively used in the treatment of type 2 diabetes mellitus (T2DM). Although both medications effectively lower plasma glucose levels, differences may exist in their pharmacokinetics and effect on the kidney. In the context of diabetic kidney disease, DPP-4 inhibitors may confer renal protection through several putative mechanisms. In contrast, sulfonylureas are associated with weight gain and cardiac dysfunction, which may adversely influence kidney function.

The investigators hypothesize that DPP-4 inhibitors and sulfonylureas may have a different effect on the diabetic kidney. This study compares the effect of DPP-4 inhibitors and sulfonylureas on urinary albumin excretion in patients with newly diagnosed T2DM.

DETAILED DESCRIPTION:
Diabetic kidney disease (DKD) occurs in a considerable number of individuals with type 2 diabetes mellitus (T2DM). DKD leads to substantial morbidity and reduces the quality of life in afflicted patients. Chronic hyperglycemia induces proapoptotic signaling pathways in mesangial cells, leading to microvascular injury in the diabetic kidney. Clinical interventions targeting plasma glucose, body weight, and blood pressure have been shown to attenuate the progression of DKD.

Dipeptidyl peptidase 4 (DPP-4) inhibitors and sulfonylureas have been extensively used in the treatment of T2DM. Although both medications effectively lower plasma glucose levels, differences may exist in their pharmacokinetics and effect on the kidney. In the context of DKD, DPP-4 inhibitors may confer renal protection through several putative mechanisms. However, whether such renal protection involves the glucose lowering efficacy of DPP-4 inhibitors or additional mechanisms remains controversial. In contrast, currently there is inadequate information concerning the effect of sulfonylureas on the development of DKD. If the glucose lowering effect of DPP-4 inhibitors is a major determinant of renal protection, then sulfonylureas may theoretically offer similar benefit by maintaining euglycemia. However, sulfonylureas are associated with weight gain and cardiac dysfunction, which may adversely influence kidney function.

Given that DPP-4 inhibitors and sulfonylureas have different effect on physiologic parameters including body weight and blood pressure, the investigators hypothesize that these medications may have different effects on the diabetic kidney. This study compares the effect of DPP-4 inhibitors and sulfonylureas on urinary albumin excretion in patients with newly diagnosed T2DM.

In this study, patients with newly diagnosed T2DM are screened for eligibility. All participants receive 1000 mg of metformin therapy at the beginning of the study. Subsequently, patients are assigned to receive either the DPP-4 inhibitor Vildagliptin 50 mg twice daily or the sulfonylurea Glimepiride 2 mg twice daily. Treatment allocation is made by a committee of endocrinologists to match participants in the treatment groups by age, body weight, serum glycated hemoglobin (HbA1c), urinary albumin-to-creatinine ratio (ACR), and serum creatinine.

At the initial clinic visit, participants receive blood tests for serum HbA1c, serum creatinine, serum alanine transferase, and plasma lipid profile after a 12-hour fast. Urine samples will be collected in the morning after a 12-hour fast, and urinary ACR is measured by the turbidimetric method. Laboratory tests for these clinical variables are repeated after 24 weeks of pharmacologic treatment. Participants who loss follow up or withdraw from the study will be assessed by an intention to treat analysis. The change in urinary ACR is defined as the primary outcome measure, whereas changes in serum HbA1c, serum creatinine, body weight, and systolic blood pressure are considered secondary outcome measures.

ELIGIBILITY:
Inclusion Criteria:

* Patients exceeding 20 years of age
* Patients with newly diagnosed type 2 diabetes mellitus
* Patients who have yet to receive antidiabetic medications

Exclusion Criteria:

* Patients with non-diabetic kidney disease
* Patients with congenital kidney abnormalities
* Patients with end stage renal disease.
* Patients who have received angiotensin-converting-enzyme inhibitor or angiotensin II receptor blocker

Ages: 20 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 101 (Actual)
Dates: Start 2016-03-01 (Actual); Primary Completion 2018-02-10 (Actual); Study Completion 2018-02-28 (Actual)

PRIMARY OUTCOMES:
Change in urinary albumin-to-creatinine ratio | 24 weeks
  Change in urinary albumin-to-creatinine ratio after pharmacologic treatment

SECONDARY OUTCOMES:
Change in serum glycated hemoglobin A1c | 24 weeks
  Change in serum glycated hemoglobin A1c after pharmacologic treatment
Change in body weight | 24 weeks
  Change in body weight after pharmacologic treatment
Change in serum creatinine | 24 weeks
  Change in serum creatinine after pharmacologic treatment
Change in systolic blood pressure | 24 weeks
  Change in systolic blood pressure after pharmacologic treatment

CONTACTS AND LOCATIONS:
Overall Officials: Shih Te Tu, MD, Study Director — Changhua Christian Hospital

IPD SHARING:
Plan to Share IPD: Yes
All individual participant data that underlie results in a publication.
Supporting Information: Study Protocol
Time Frame: Starting immediately after publication.
Access Criteria: Available to any interested researcher.

REFERENCES:
- [Background] Park CW. Diabetic kidney disease: from epidemiology to clinical perspectives. Diabetes Metab J. 2014 Aug;38(4):252-60. doi: 10.4093/dmj.2014.38.4.252. PMID 25215271
- [Background] Stanton RC. Clinical challenges in diagnosis and management of diabetic kidney disease. Am J Kidney Dis. 2014 Feb;63(2 Suppl 2):S3-21. doi: 10.1053/j.ajkd.2013.10.050. PMID 24461728
- [Background] Mishra R, Emancipator SN, Kern T, Simonson MS. High glucose evokes an intrinsic proapoptotic signaling pathway in mesangial cells. Kidney Int. 2005 Jan;67(1):82-93. doi: 10.1111/j.1523-1755.2005.00058.x. PMID 15610231
- [Background] Kim MK. Treatment of diabetic kidney disease: current and future targets. Korean J Intern Med. 2017 Jul;32(4):622-630. doi: 10.3904/kjim.2016.219. Epub 2017 Jun 30. PMID 28704915
- [Background] Introduction: Standards of Medical Care in Diabetes-2018. Diabetes Care. 2018 Jan;41(Suppl 1):S1-S2. doi: 10.2337/dc18-Sint01. No abstract available. PMID 29222369
- [Background] Davidson JA. The placement of DPP-4 inhibitors in clinical practice recommendations for the treatment of type 2 diabetes. Endocr Pract. 2013 Nov-Dec;19(6):1050-61. doi: 10.4158/EP12303.RA. PMID 24126227
- [Background] Makino Y, Fujita Y, Haneda M. Dipeptidyl peptidase-4 inhibitors in progressive kidney disease. Curr Opin Nephrol Hypertens. 2015 Jan;24(1):67-73. doi: 10.1097/MNH.0000000000000080. PMID 25415611
- [Background] Sola D, Rossi L, Schianca GP, Maffioli P, Bigliocca M, Mella R, Corliano F, Fra GP, Bartoli E, Derosa G. Sulfonylureas and their use in clinical practice. Arch Med Sci. 2015 Aug 12;11(4):840-8. doi: 10.5114/aoms.2015.53304. Epub 2015 Aug 11. PMID 26322096